CLINICAL TRIAL: NCT04911959
Title: Study on the Safety and Effectiveness of Transcatheter Arterial Chemoembolization (TACE) Combined With Lenvatinib to Prevent Postoperative Recurrence in Patients With Microvascular Invasion (MVI) Positive Hepatocellular Carcinoma (HCC)
Brief Title: Study of TACE Combined With Lenvatinib to Prevent Postoperative Recurrence in Patients With MVI Positive HCC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: yan2020-629
Record Dates: First submitted 2021-01-18; First posted 2021-06-03 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma; Lenvatinib
Keywords: TACE; Hepatocellular Carcinoma; MVI; Prognosis; Lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): patients receive transcatheter arterial chemoembolization (TACE) only.
  Interventions: Procedure: TACE
- Intervention group (Experimental): patients receive transcatheter arterial chemoembolization (TACE) and lenvatinib 8mg per day.
  Interventions: Drug: Lenvatinib; Procedure: TACE

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib is taken orally.
  Arms: Intervention group
Procedure: TACE — TACE treatment once.
  Other Names: Transcatheter Arterial Chemoembolization

SUMMARY:
single-center clinical trial studies have verified the safety and effectiveness of transcatheter arterial chemoembolization (TACE) combined with lenvatinib in preventing postoperative recurrence of microvascular invasion (MVI) positive HCC patients. Explore a new clinical first-line treatment plan for patients with liver cancer microvascular invasion after surgery.

DETAILED DESCRIPTION:
Focusing on the current status of clinical treatment of microvascular invasion (MVI) positive postoperative hepatocellular carcinoma (HCC) , single-center clinical trial studies have verified the safety and effectiveness of transcatheter arterial chemoembolization (TACE) combined with lenvatinib in preventing postoperative recurrence of MVI-positive HCC patients. Explore a new clinical first-line treatment plan for patients with liver cancer microvascular invasion after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Radical hepatocellular carcinoma was treated 4 weeks (±1 week) ago, and the pathological diagnosis was HCC after surgery, and MVI was positive
* Child-Pugh score ≤9 points (Child-Pugh A-B), PS score 0-2 points, BCLC stage A-B
* The main portal vein is not completely obstructed, or although it is completely obstructed, the compensatory collateral branches of the portal vein are abundant or the portal vein blood flow can be restored by implanting the portal vein stent
* With sufficient organ and bone marrow function, the laboratory test values within 7 days before enrollment meet the requirements
* Physical fitness score ECOG 0～2
* Expected survival> 3 months
* No other systemic malignancies
* Female subjects of childbearing age or male subjects whose sexual partners are females of childbearing age must take effective contraceptive measures throughout the treatment period and 6 months after the treatment period
* Subjects have informed consent, understand and are willing to cooperate with the trial protocol, and sign relevant documents

Exclusion Criteria:

* Histology includes fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma, etc.
* Severe liver dysfunction (Child-Pugh C), including jaundice, hepatic encephalopathy, refractory ascites, hepatorenal syndrome, or a history of liver transplantation
* The main portal vein is completely blocked, and the formation of collateral vessels is small

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 8 weeks
  To evaluate the safety of TACE combined with lenvatinib treatment in preventing postoperative recurrence in patients with MVI-positive HCC
Changes in tumor volume | Up to 8 weeks
  To evaluate the effectiveness of TACE combined with lenvatinib treatment in preventing postoperative recurrence in patients with MVI-positive HCC
Recurrence-free survival (RFS) evaluation | Through study completion, an average of 1 year
  To evaluate the recurrence-free survival of patients with MVI-positive HCC after TACE combined with lenvatinib treatment

SECONDARY OUTCOMES:
Disease recurrence time evaluation | Through study completion, an average of 1 year
  To evaluate the tumor recurrence time of patients with MVI-positive HCC after TACE combined with lenvatinib treatment
Overall survival ( OS) evaluation | Through study completion, an average of 1 year
  Overall survival time as assessed by IRC

CONTACTS AND LOCATIONS:
Overall Officials: Zhongquan Sun, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (2):
- China (2):
  - Weilin Wang, Hangzhou, None Selected
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang